CLINICAL TRIAL: NCT01263600
Title: Cohort Hepatitis B Virus (HBV) Pediatric Protocol
Brief Title: Hepatitis B Research Network Pediatric Cohort Study (HBRN)
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Anna Lok, Study Chair, University of Michigan
Other Study IDs: DK082864Pediatric; U01DK082916 (NIH); U01DK082864 (NIH); U01DK082874 (NIH); U01DK082944 (NIH); U01DK082843 (NIH); U01DK082871 (NIH); UL1TR000423 (NIH); UL1TR000004 (NIH); A-DK-3002-001 (Other: Interagency Agreement)
Record Dates: First submitted 2010-12-14; First posted 2010-12-20 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; HBV; Pediatric
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsy tissue, blood (serum, plasma, and DNA)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to describe participants 6 months to <18 years of age with hepatitis B virus (HBV) infection in a prospective cohort in the United States (US) and Canada and identify predictors of disease activation and progression.

DETAILED DESCRIPTION:
•Primary Aim:

o To describe participants 6 months to <18 years of age with hepatitis B virus (HBV) infection in a prospective cohort in the United States (US) and Canada and identify predictors of disease activation and progression

Secondary Aims:

* To describe clinical, virological, and immunological characteristics of participants with HBV in the US and Canada.
* To evaluate changes in HBV infection status and hepatitis B surface antigen (HBsAg) levels and factors associated with those changes.
* To verify whether a baseline HBsAg below 1,000 IU/mL and HBV DNA below 1,000 IU/mL is an accurate predictor of people who are, or who will become, inactive carriers, defined as people who are HBsAg positive, hepatitis B "e" antigen (HBeAg) negative, have normal alanine aminotransferase (ALT) and HBV DNA under 1,000 IU/mL on at least two occasions over a period of at least 6 months with HBV DNA under 1,000 IU/mL.
* To assess the health related quality of life (HRQOL) of treatment naïve hepatitis B surface antigen (HBsAg) positive children and adolescents
* To develop a bank of biospecimens (e.g., serum, plasma, DNA, liver tissue) obtained from participants with HBV infection.
* To identify pediatric participants from 2 years to <18 years of age with chronic HBV infection for potential participation in treatment study to be conducted by the Hepatitis B Research Network (HBRN).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent as appropriate
* At least 6 months to <18 years of age
* Hepatitis B surface antigen (HBsAg) positive

Exclusion Criteria:

* Hepatic decompensation
* Hepatocellular carcinoma (HCC)
* Liver transplantation
* Current Hepatitis B antiviral treatment (except pregnant females)
* Known coinfection with HIV (patients with hepatitis D or hepatitis C coinfection are not excluded)
* Medical or social condition which in the opinion of the principal investigator would interfere with or prevent regular follow up.
* Unable or unwilling to return for regular follow-up

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients from Children's Hospitals and university medical centers in the United States and Canada
Sampling Method: Non-Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2010-12; Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Antigen loss: e and s | up to 288 weeks
  Loss of these viral markers may be associated with appearance of corresponding antibodies in serum (anti-HBe or anti-HBs). HBsAg loss appears to represent a "cure" of HBV infection and is associated with reduction, but not necessarily elimination, of the risk of future complications, such as Hepatocellular carcinoma (HCC) which may occur, particularly in those who lose HBsAg at an older age (after 50 years) or after the development of cirrhosis. When HBeAg or HBsAg loss occurs, participants will be followed more closely initially and then return to the regular follow-up schedule.

SECONDARY OUTCOMES:
Hepatitis exacerbation marked by alanine aminotransferase (ALT) Flare | up to 288 weeks
  A flare is defined as serum alanine aminotransferase (ALT) greater than or equal to 10 times the upper limit of normal which corresponds to (1 550 IU/L in females and 600 IU/L in males for 6 months - 18 months of age and 2) 350 IU/L in females and 400 IU/L in males for >18 months - < 18 years of age (12). Once a flare is detected, participants will be followed more closely until its resolution.
Cirrhosis | up to 288 weeks
  The diagnosis of cirrhosis will be made by (1) liver histology, when available or In the absence of histological diagnosis, cirrhosis is defined as any one of the following
  * Presence of ascites or hepatic hydrothorax
  * Variceal or portal hypertensive bleeding
  * Hepatic encephalopathy
  * Child-Turcotte-Pugh (CTP) score of 7 or above
  or in the absence of hepatic decompensation (any two of the following):
  * Splenomegaly
  * Nodular liver
  * Platelet count below 120,000/mm3
  Once cirrhosis is diagnosed, patient follow-up should include Hepatocellular carcinoma(HCC)surveillance
Hepatic Decompensation | up to 288 weeks
  It is likely that the development of cirrhosis and subsequent hepatic decompensation will be preceded and foreseen by the progression of fibrosis. Development of hepatic decompensation will be defined by any of the following events:
  * Ascites or hepatic hydrothorax
  * Variceal bleeding or portal hypertensive bleeding
  * Hepatic encephalopathy
  * Child-Turcotte-Pugh (CTP) score of 7 or above
  It is anticipated that there will be a small number of patients that will develop decompensation during the follow-up.
Hepatocellular carcinoma (HCC) | up to 288 weeks
  HCC may be detected by routine surveillance or may become clinically apparent. The diagnosis of HCC will be made using the American Association for the Study of Liver Disease criteria.
Death | up to 288 weeks
  Death may occur related to liver disease (typically hepatic decompensation or HCC) or may occur unrelated to hepatitis B or liver disease. Date and cause of death will be recorded.
Liver transplantation | up to 288 weeks
  Liver transplantation will be recorded upon notification. Date of transplantation, indication for transplantation, and occurrence of incidental HCC will be recorded. Follow-up ends with liver transplantation.
Reaching 18 years of Age | up to 288 weeks
  Patients who reach 18 years of age and are within an adult HBRN clinical center will be offered participation in the adult cohort study and re-consented for the adult protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Belle, PhD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (6):
  - University of California San Francisco Medical Center, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - University of Texas Southwestern, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Bisceglie AM, King WC, Lisker-Melman M, Khalili M, Belle SH, Feld JJ, Ghany MG, Janssen HLA, Lau D, Lee WM, Ling SC, Cooper S, Rosenthal P, Schwarz KB, Sterling RK, Teckman JH, Terrault N; Hepatitis B Research Network (HBRN). Age, race and viral genotype are associated with the prevalence of hepatitis B e antigen in children and adults with chronic hepatitis B. J Viral Hepat. 2019 Jul;26(7):856-865. doi: 10.1111/jvh.13104. Epub 2019 May 2. PMID 30974509
- See also: The Hepatitis B Research Network study web site — http://www.hepbnet.org/